CLINICAL TRIAL: NCT01218633
Title: A Dose-response Study of the Effects of Exendin-9,39 on Glucose Metabolism, Glucagon and Insulin Secretion and on Insulin Action.
Brief Title: Dose-response Study of Exendin-9,39 on Glucose Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adrian Vella (Other)
Responsible Party: Sponsor-Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10-003435
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Effects of 9,39-Exendin and 9,36-GLP-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline (Placebo Comparator)
  Interventions: Drug: saline infusion
- GLP-1-(9,36)-amide (Active Comparator)
  Interventions: Drug: GLP-1-9,36 infusion
- Exendin-9,39 @30pmol/kg/min (Active Comparator)
  Interventions: Drug: Exendin-9,39 at low dose
- Exendin-9,39 @300pmol/kg/min (Active Comparator)
  Interventions: Drug: Exendin-9,39 at high dose

INTERVENTIONS:
Drug: saline infusion — saline infused at 30ml/hour
  Arms: Saline
Drug: GLP-1-9,36 infusion — infused @ 1.2pmol/kg/min
  Arms: GLP-1-(9,36)-amide
Drug: Exendin-9,39 at low dose — infused at 30pmol/kg/min
  Arms: Exendin-9,39 @30pmol/kg/min
Drug: Exendin-9,39 at high dose — infused @ 300pmol/kg/min
  Arms: Exendin-9,39 @300pmol/kg/min

SUMMARY:
Multiple studies have examined the effect of endogenous GLP-1 secretions by using a competitive antagonist of GLP-1 - Exendin-9,39 - infused at rates of 300pmol/kg/min. However, the presence of an effect does not necessarily imply that this effect is due to the blockade of the endogenous GLP-1 actions at the receptor. It is possible that the supraphysiologic concentrations of Exendin may have effects of its own. To examine the effect of Exendin on glucose metabolism the investigators propose a dose-response study to determine whether the compound has effects in a dose-dependent fashion.

ELIGIBILITY:
Healthy Not on any medication other than thyroid hormone replacement or OCP No history of diabetes No prior upper GI surgery

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Insulin Secretion | over 360 minutes of study

SECONDARY OUTCOMES:
glucagon secretion | over 360 minutes of study

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Sathananthan M, Farrugia LP, Miles JM, Piccinini F, Dalla Man C, Zinsmeister AR, Cobelli C, Rizza RA, Vella A. Direct effects of exendin-(9,39) and GLP-1-(9,36)amide on insulin action, beta-cell function, and glucose metabolism in nondiabetic subjects. Diabetes. 2013 Aug;62(8):2752-6. doi: 10.2337/db13-0140. Epub 2013 Apr 1. PMID 23545708